CLINICAL TRIAL: NCT01383473
Title: Concurrent School Attendance And Cancer Therapy: The Experiences of 6-12 Year Old Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCHOOL1
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia; Lymphoma; Solid Tumor
Keywords: cancer therapy; school attendance; cancer diagnosis; perception
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Leukemia Patients: 6-12 year old pediatric oncology patients' perceptions of their school experiences pre and post cancer diagnosis will be done through interviews and drawings.
- Solid Tumor Patients: 6-12 year old pediatric oncology patients' perceptions of their school experiences pre and post cancer diagnosis will be done through interviews and drawings.

SUMMARY:
Many children with cancer cannot participate regularly in school due to frequent hospitalizations for treatment or treatment related effects such as pain, nausea, and fatigue. Prior studies have shown that children with cancer desire to attend school while receiving therapy despite these challenges, and that they report psychological and psychosocial difficulties if unable to attend. While school attendance has been found to correlate with Health-Related Quality of Life (HRQoL), self-efficacy beliefs, and self-esteem, little is known about how children with cancer experience school attendance while receiving active cancer therapy. The purpose of this study will be to explore how 6-12 year old children with cancer perceive school attendance pre and post diagnosis during active therapy as measured at one-time point, 6 months (± 2months) into active therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to explore 6-12 year old pediatric oncology patients' perceptions of their school experiences pre and post cancer diagnosis.

This study will utilize qualitative interview methods. Potential participants who meet inclusion criteria will be approached by the principal investigator to obtain consent and assent in accordance with institutional guidelines. Upon giving consent, the child will participate in a one-hour audio-taped interview session with the principal investigator. The interview session will begin with some general rapport building questions to help the child grow comfortable with the interviewer, the interview room, and the interview format. The rest of the interview will consist of questions pertaining to the child's school experiences both before and during diagnosis and treatment for malignancy. The interview will conclude with the child being asked to draw a picture of themselves at school before diagnosis, and of themselves at school since being diagnosed. Demographic data will be collected from each participant's medical chart pertaining to age, gender, ethnicity, diagnosis, and the type of school attended before and after diagnosis and the principal investigator and study staff involved in data coding will complete field note entries directly following the conclusion of each interview or data coding session (see Appendix V). The participant's involvement in the study will end at the conclusion of the interview session.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 6-12 years of age at the time of diagnosis.
* Participant has a primary diagnosis of leukemia/lymphoma or solid tumor.
* Participant has been on therapy for six months (plus or minus 2 months) at the time of enrollment on this protocol.
* Participant is able to read and speak English.

Exclusion Criteria:

* Participant has not received any type of schooling services either in the home, community, or hospital setting since diagnosis.
* Participant did not receive any type of schooling services prior to diagnosis.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will consist of 6-12-year-old patients currently on therapy for a primary diagnosis of a leukemia/lymphoma or solid tumor at St. Jude Children's Research Hospital in Memphis, Tennessee. Potential participants will be recruited via a medical chart review performed by the principal investigator in order to identify children who have been on active therapy for a malignancy for 6 months (plus or minus 2 months) at the time of enrollment on this protocol
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
6-12 year old pediatric oncology patients' perceptions of their school experiences pre and post cancer diagnosis will be explored; | 1 year
  This will be done through interviews and drawings.

CONTACTS AND LOCATIONS:
Overall Officials: Jessika C Boles, MEd., CCLS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org